CLINICAL TRIAL: NCT04689724
Title: Determining Airway Management Related Outcomes in COVID19 Patients and in Health Care Providers
Brief Title: Covid-19 Airway Management
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Matteo Parotto, Dr. Matteo Parotto, University Health Network, Toronto
Other Study IDs: 20-5620
Record Dates: First submitted 2020-12-29; First posted 2020-12-30 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Covid-19_airways Management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study has a retrospective and a prospective component. The retrospective component aims to review data of all airway management related SAEs in COVID 19 patients (between April and July 2020); hypoxemia, hypotension and cardiac arrest within 15 min of intubation. The prospective component aims to assess the incidence of COVID-19 infection in Airway Management Team members by means of an interview assessing their COVID19 status after participating in airway management in the period outlined above. This prospective interview component is starting in December 2020.

DETAILED DESCRIPTION:
Approximately 5-10% of all patients affected by COVID-19 develop severe respiratory distress. This has already involved hundreds of people in Ontario and thousands worldwide. In this situation, support with a mechanical ventilator is required. The first essential step to provide this support is to insert a breathing tube in the patent's trachea (windpipe), a process called 'endotracheal intubation' or more broadly, 'airway management'. While a fundamental lifesaving resource, endotracheal intubation in COVID-19 patents is a highly specialized procedure that carries risk both to patents and attending healthcare providers as follows. a) Clinicians involved in airway management for patients with coronaviruses are at extremely high risk of infection due to aerosol and droplet exposure during the procedure. b) Rapid administration of drugs that put the patent to sleep is usually required for prompt and safe endotracheal intubation. However, in physiologically compromised patents, life-threatening side-effects may occur, such as very low oxygen levels (in as many as 70% of patients), low blood pressure (18-22% of patients), and cardiac arrest (2%); these can significantly affect outcomes. No definitive data are presently available to accurately quantify the risk posed by such procedures to healthcare professionals and patents, nor the associated factors. We have developed a retrospective study reviewing data all airway management related SAEs in COVID 19 patients (between April and July 2020); hypoxemia, hypotension and cardiac arrest within 15 min of intubation. Additionally, we are going to prospectively interview Airway Management Team members that were involved in the airway management of COVID19 patients in the period described above, in order to assess whether they developed signs and symptoms and/or a confirmed COVID19 infection. This prospective interview component is starting in December 2020.

ELIGIBILITY:
Inclusion Criteria:

All Suspected or confirmed Covid-19 patients that require intubation Health care workers from the airways management team who performed an intubation on confirmed or suspected Covid-19 patients

Exclusion Criteria:

Lack of Health Care Provider Consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will use exclusively retrospective data from suspected or positive COVID-19 adult patients who required intubation during their hospital stay and also record the rate of infection in HCP who perform the intubation.
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2021-10-27 (Actual)

PRIMARY OUTCOMES:
Serious adverse events at intubation | within 15 min of intubation
  hypoxemia, hypotension and cardiac arrest within 15 min of intubation in confirmed or suspected COVID-19 patients

SECONDARY OUTCOMES:
Signs, symptoms or confirmed COVID19 infection in healthcare providers | within 14 days after participating in airway management for confirmed or suspected COVID-19 patients
  via an interview exploring past events, we will assess whether providers recall having developed signs, symptoms or confirmed COVID19 infection after participating in airway management for confirmed or suspected COVID-19 patients

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Parotto, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Result] Jarvis N, Schiavo S, Bartoszko J, Ma M, Chin KJ, Parotto M. A specialized airway management team for COVID-19 patients: a retrospective study of the experience of two Canadian hospitals in Toronto. Can J Anaesth. 2022 Mar;69(3):333-342. doi: 10.1007/s12630-021-02169-x. Epub 2021 Dec 8. PMID 34881407